CLINICAL TRIAL: NCT02754440
Title: Evaluation of the Performance of Trima Accel® Version 7.0 Software Enhancements for the Collection of Platelets Stored in Platelet Additive Solution
Brief Title: Evaluation of Trima Version 7.0 Platelets in PAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Terumo BCT (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CTS-5059
Record Dates: First submitted 2016-04-26; First posted 2016-04-28 (Estimated); Results first posted 2018-05-11 (Actual); Last update posted 2018-05-11 (Actual); Status verified 2018-04

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Single Platelet Product (Experimental): Healthy adult volunteer blood donors that qualify for a single unit platelet collection will undergo plateletpheresis on the Trima Accel® Automated Blood Collection System (Trima Accel System with Version 7.0 Software). Concurrent plasma will be collected in 25% of the collections.
  Interventions: Device: Trima Accel System with Version 7.0 Software
- Double Platelet Product (Experimental): Healthy adult volunteer blood donors that qualify for a double unit platelet collection will undergo plateletpheresis on the Trima Accel® Automated Blood Collection System (Trima Accel System with Version 7.0 Software). Concurrent plasma will be collected in 25% of the collections.
  Interventions: Device: Trima Accel System with Version 7.0 Software
- Triple Platelet Product (Experimental): Healthy adult volunteer blood donors that qualify for a triple unit platelet collection will undergo plateletpheresis on the Trima Accel® Automated Blood Collection System (Trima Accel System with Version 7.0 Software). Concurrent plasma will be collected in 25% of the collections.
  Interventions: Device: Trima Accel System with Version 7.0 Software

INTERVENTIONS:
Device: Trima Accel System with Version 7.0 Software — Platelet Apheresis Procedure

SUMMARY:
To verify that platelets collected on the Trima Accel system with Version 7.0 software enhancements and stored in platelet additive solution (PAS) meet the FDA requirements for leukoreduction (< 5.0 × 10^6 residual white blood cells [WBC] per transfusable unit).

DETAILED DESCRIPTION:
The study is designed to evaluate changes to the Trima Accel software to ensure the modified software meets the FDA acceptance criteria for leukoreduction and platelet yield. The operating range for the system flow rates, anticoagulant ratios, storage conditions, and centrifugal forces are the same as the currently cleared Trima Accel system. There are no changes to the environment or storage conditions for platelets, therefore, no in vitro or in vivo platelet quality data will be collected.

This is a prospective, open-label, multi-center controlled study to evaluate the leukoreduction of platelets stored in platelet additive solution (PAS) collected on the Trima Accel system Version 7.0 software enhancement. Up to 450 healthy adult subjects will be enrolled in this study to ensure 93 single, 93 double and 93 triple platelet product evaluable data points. Evaluable is defined as a completed platelet product that does not meet any of the protocol analysis exclusion criteria.

Plateletpheresis will be per site standard practice and per applicable FDA guidelines such as the FDA Collection of Platelets by Automated Methods, December 2007 Guidance for Industry and Pre-storage Leukocyte Reduction of Whole Blood and Blood Components Intended for Transfusion, September 2012.

Study participation will be up to 30 days and will consist of 1 to 2 visits. Screening may be done within 30 days before the apheresis procedure or combined as a single visit, which includes screening and the apheresis procedure all in 1 day.

The entire study should be completed in approximately 16 months.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older.
* Meets the inclusion criteria defined by the Blood Center for an apheresis platelet with PAS collection on the Trima Accel system. These criteria are based on FDA guidance and American Association of Blood Banks (AABB) standards. Note: subjects who are deferred from volunteer community donations because of travel restrictions, piercings, or tattoos may participate in the study, as products are not transfused.
* Has given written informed consent.

Exclusion Criteria:

* Has previously donated an evaluable platelet product in this study (CTS 5059).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 365 (Actual)
Dates: Start 2016-04-20 (Actual); Primary Completion 2017-07-28 (Actual); Study Completion 2017-07-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heather Pidcoke, MD, PhD, Study Director — Terumo BCT, Inc
Locations (7):
- United States (7):
  - San Diego Blood Bank, San Diego, California
  - Bonfils Blood Center, Denver, Colorado
  - Indiana Blood Center, Indianapolis, Indiana
  - Memorial Blood Centers, Minneapolis, Minnesota
  - Community Blood Center of Greater Kansas, Kansas City, Missouri
  - Hoxworth Blood Center, Cincinnati, Ohio
  - Blood Center of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A participant was considered "enrolled" upon signing the informed consent form.
Pre-assignment Details: 365 participants consented/enrolled: 25 screen-failed; 5 never started procedure = 30 participants excluded from Safety Analysis.
  335 participants = Safety Analysis set (56 participants excluded from the full analysis set: 35 participants were "unassigned" to an Arm, 21 participants were assigned to an Arm)
  279 = Full Analysis set
Groups:
- Unassigned: Participant and subsequent platelet product not assignable as single, double, triple (product not tested and/or was excluded from analysis).
Period: Overall Study
Arm/Group | Single Platelet Product | Double Platelet Product | Triple Platelet Product | Unassigned
Started | 99 | 101 | 100 | 35
Completed | 93 | 93 | 93 | 0
Not Completed | 6 | 8 | 7 | 35
Not completed — Protocol Violation | 3 | 2 | 2 | 6
Not completed — Adverse Event | 3 | 1 | 0 | 9
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1
Not completed — Equipment failure | 0 | 5 | 5 | 7
Not completed — Subject issues not resulting in AE | 0 | 0 | 0 | 12

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set = Includes all Subjects that had an apheresis procedure started.
Groups:
- Total: Total of all reporting groups
Arm/Group | Single Platelet Product | Double Platelet Product | Triple Platelet Product | Unassigned | Total
Number analyzed (Participants) | 99 | 101 | 100 | 35 | 335
Age, Customized [Count of Participants; unit: Participants]
  Age ≥ 18 years | 99 | 101 | 100 | 35 | 335
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 43 | 43 | 17 | 146
  Male | 56 | 58 | 57 | 18 | 189
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 2 | 2 | 0 | 5
  Black | 2 | 3 | 3 | 2 | 10
  Hispanic | 1 | 7 | 6 | 1 | 15
  White | 93 | 86 | 84 | 28 | 291
  No Response | 0 | 1 | 2 | 1 | 4
  Unknown | 1 | 2 | 0 | 2 | 5
  Other | 1 | 0 | 3 | 1 | 5
Region of Enrollment [Number; unit: participants]
  United States | 99 | 101 | 100 | 35 | 335
Height [Mean (Standard Deviation); unit: inches] | 68.6 (3.90) | 68.7 (3.95) | 69.1 (4.04) | 69.5 (4.28) | 68.9 (3.99)
Weight [Mean (Standard Deviation); unit: pounds] | 202.25 (42.04) | 205.09 (46.95) | 225.01 (51.3) | 207.45 (51.44) | 210.44 (48.18)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Platelet Units Containing an Acceptable Residual WBC Level
Description: The number of participants with platelet units containing an acceptable residual WBC level. Acceptable residual WBC counts are: singles = residual WBC level < 5.0 × 10^6; doubles = residual WBC level < 8.0 × 10^6 or < 5.0 × 10^6 for each transfusable unit; and triples = residual WBC level < 12.0 × 10^6 or < 5.0 × 10^6 for each transfusable unit.
Time Frame: Within 48 hours of end of donation
Population: The Full Analysis Set (FAS) included all participants that completed the study and did not meet any of the protocol exclusion criteria. A participant could only have 1 product included in the FAS. The FAS was used to examine the primary and secondary endpoints.
Measure: Count of Participants; unit: Participants
Arm/Group | Single Platelet Product | Double Platelet Product | Triple Platelet Product
Number analyzed (Participants) | 93 | 93 | 93
Participants
  Success (N) | 93 | 93 | 93
  Failure (N) | 0 | 0 | 0
Statistical Analysis 1: Comparison: Single Platelet Product; Up to 450 healthy adult subjects will be enrolled in this study to ensure 93 evaluable single platelet product collections, 93 evaluable double platelet product collections, and 93 evaluable triple platelet product collections. This number was chosen to meet the FDA requirements of at least 95% of platelet units with an acceptable residual WBC level with 95% confidence. With 93 platelet products, this allowed for at most 1 failure; Test type: Other — A procedure is a success if the subject's platelet product has a residual WBC count of < 5.0 × 10^6 for the single platelet product group. The FDA requirements are met if the lower one-sided 95% confidence interval for the procedure success rate is at least 95%; Simple Sample Proportion = 1.00, 95% CI 1-sided [lower limit 0.968], Standard Error of Mean 0 — When estimated proportion is 100%, standard error of the mean is estimated as 0
Statistical Analysis 2: Comparison: Double Platelet Product; [analysis description as in outcome 1, analysis 1]; Test type: Other — A procedure is a success if the subject's platelet product has a residual WBC count of < 8.0 × 10^6 for the double platelet product group, or < 5.0 × 10^6 for each transfusable unit . The FDA requirements are met if the lower one-sided 95% confidence interval for the procedure success rate is at least 95%; Simple Sample Proportion = 1.00, 95% CI 1-sided [lower limit 0.968], Standard Error of Mean 0 — When estimated proportion is 100%, standard error of the mean is estimated as 0
Statistical Analysis 3: Comparison: Triple Platelet Product; [analysis description as in outcome 1, analysis 1]; Test type: Other — A procedure is a success if the subject's platelet product has a residual WBC count of < 12.0 × 10^6 for the triple platelet product group, or < 5.0 × 10^6 for each transfusable unit . The FDA requirements are met if the lower one-sided 95% confidence interval for the procedure success rate is at least 95%; Simple Sample Proportion = 1.00, 95% CI 1-sided [lower limit 0.968], Standard Error of Mean 0 — When estimated proportion is 100%, standard error of the mean is estimated as 0

2. Secondary Outcome: Number of Participants With Platelet Units Containing an Acceptable Platelet Yield
Description: The number of participants with platelet units containing an acceptable platelet yield. Acceptable platelet yield for single, double and triple platelet products are: platelet yield ≥ 3.0 × 10^11 for singles, platelet yield ≥ 6.2 × 10^11 for doubles, and platelet yield ≥ 9.3 × 10^11 for triples.
Time Frame: Within 48 hours of end of donation
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Single Platelet Product | Double Platelet Product | Triple Platelet Product
Number analyzed (Participants) | 93 | 93 | 93
Participants
  Success (N) | 89 | 93 | 93
  Failure (N) | 4 | 0 | 0
Statistical Analysis 1: Comparison: Single Platelet Product; Up to 450 healthy subjects were enrolled to ensure 93 evaluable single, double, and triple platelet product collections. With 93 platelet products being collected, 16 failures or less was required to show that the proportion of units with an acceptable platelet yield is at least 75% with 95% confidence; Test type: Other — A procedure is a success if the subject's platelet product has a platelet yield of ≥ 3.0 × 10^11 for the single platelet product group. The requirements are met if the lower one-sided 95% confidence interval for the procedure success rate is at least 75%; Simple Sample Proportion = 0.957, 95% CI 1-sided [lower limit 0.904], Standard Error of Mean 0.0210
Statistical Analysis 2: Comparison: Double Platelet Product; [analysis description as in outcome 2, analysis 1]; Test type: Other — A procedure is a success if the subject's platelet product has a platelet yield of ≥ 6.2 × 10^11 for the double platelet product group. The requirements are met if the lower one-sided 95% confidence interval for the procedure success rate is at least 75%; Simple Sample Proportion = 1.00, 95% CI 1-sided [lower limit 0.968], Standard Error of Mean 0 — When estimated proportion is 100%, standard error of the mean is estimated as 0
Statistical Analysis 3: Comparison: Triple Platelet Product; [analysis description as in outcome 2, analysis 1]; Test type: Other — A procedure is a success if the subject's platelet product has a platelet yield of ≥ 9.3 × 10^11 for the triple platelet product group. The requirements are met if the lower one-sided 95% confidence interval for the procedure success rate is at least 75%; Simple Sample Proportion = 1.00, 95% CI 1-sided [lower limit 0.968], Standard Error of Mean 0 — When estimated proportion is 100%, standard error of the mean is estimated as 0

ADVERSE EVENTS:
Time Frame: Adverse events that occurred from the time of signing informed consent, through the screening period of up to 30 days, and on the day of the apheresis procedure were recorded. On the day of the apheresis procedure, adverse event monitoring stopped at the time participants left the blood center, which was considered study completion.
Description: Treatment emergent adverse events were analyzed in the Safety Analysis set. Treatment begin with the apheresis venipuncture
Arm/Group | Single Platelet Product | Double Platelet Product | Triple Platelet Product | Unassigned
All-Cause Mortality (participants affected / at risk) | 0/99 | 0/101 | 0/100 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/99 | 0/101 | 0/100 | 0/35
Other Adverse Events (participants affected / at risk) | 10/99 | 8/101 | 9/100 | 10/35
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Platelet Product (N=99) | Double Platelet Product (N=101) | Triple Platelet Product (N=100) | Unassigned (N=35)
Citrate Toxicity (Metabolism and nutrition disorders) | 10 (10) | 8 (8) | 9 (9) | 0 (0)
Hematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 8 (8)
Injection Site Extravasation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor retains the right to review and comment on any public disclosure of study results. If no response is received within 30 days, the Principal Investigator may presume that the submission for publication may proceed without delay. If the Sponsor asks to defer publication, Study Site shall not publish, or otherwise disclose to any third party, any of the information contained in the publication or presentation until such time as permission is granted from the Sponsor.

DOCUMENTS (3):
  • Study Protocol (2016-11-22): https://cdn.clinicaltrials.gov/large-docs/40/NCT02754440/Prot_000.pdf
  • Informed Consent Form (2016-11-22): https://cdn.clinicaltrials.gov/large-docs/40/NCT02754440/ICF_001.pdf
  • Statistical Analysis Plan (2017-05-17): https://cdn.clinicaltrials.gov/large-docs/40/NCT02754440/SAP_002.pdf